CLINICAL TRIAL: NCT05874960
Title: Helicobacter Pylori Prevalence in Southern Region of Romania
Acronym: HELIUM
Status: Completed | Type: Observational
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Mihai Ciocirlan, Associate Professor, Carol Davila University of Medicine and Pharmacy
Other Study IDs: HELIUM
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Infections, Helicobacter
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study, voluntary participation, 12 months, studying Helicobacter pylori prevalence.

DETAILED DESCRIPTION:
Observational study, voluntary participation, 12 months, studying Helicobacter pylori prevalence.

The aim of the study is to evaluate the prevalence of H. pylori infection in several areas of the Southern Regions of Romania, considered as vulnerable pertaining to the access of health services.

Fecal Helicobacter pylori will be tested, together with antibiotic susceptibility.

ELIGIBILITY:
Inclusion Criteria:

* Adult voluntary participants to "Medical services caravan" project by Medcorp Association

Exclusion Criteria:

* Age < 18 years old
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult population from Southern Regions of Romania, from rural vulnerable areas concerning access to health services.
Sampling Method: Non-Probability Sample
Enrollment: 708 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori infection rate | 12 months
  rate of fecal antigen test divided by total number of tests (fecal Helicobacter test)

SECONDARY OUTCOMES:
Antibiotic susceptibility rate | 12 months
  rate of antibiotic (x) susceptibility divided by total number of tests (antibiotic susceptibility test)

CONTACTS AND LOCATIONS:
Overall Officials: Radu Prodan, MD, Principal Investigator — Medcorp Association
Locations (1):
- Medcorp Association, Bucharest, Romania